CLINICAL TRIAL: NCT03148821
Title: Pressure Area Distribution on a Variety of Clinical Surfaces in a Group of 51 Volunteers
Brief Title: Pressure Area Distribution on a Variety of Clinical Surfaces
Status: Withdrawn | Type: Observational
Why Stopped: Loss of promised funding
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 169214
Record Dates: First submitted 2017-04-06; First posted 2017-05-11 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Pressure Ulcer
Keywords: pressure ulcer; pressure sore; patient positioning
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteer participants: The investigators propose a snap shot study in a group of healthy volunteers of varying BMIs, laying on surfaces a patient would be exposed to during their hospital stay. Participants will lie on a variety of surfaces they may find themselves on during an emergency admission to hospital, including an operating table, in a variety of positions. Participants pressure distributions in each scenario will be measured with a pressure sensing mattress.

SUMMARY:
Participants in the study will be adults with full mobility, with the capacity to give informed written consent. The investigators will recruit a group of volunteers in order to represent a variety of BMIs, in an attempt to gain a sample of the BMIs found in the population. The investigators will mimic current practices and standard equipment in order to replicate real conditions as closely as possible.

Participants will lay on the following surfaces in the following scenarios

1. Ambulance scoop: supine (lying flat on their back)
2. A&E trolley: supine
3. Hospital bed: supine
4. Theatre table: supine
5. Theatre table: Left lateral (lying on their left side at 90 degrees to the operating table) with pelvic binders (pads designed to keep the hip immobile).

Each participant will remain in each position on that particular surface for a period of 25 minutes. A pressure mapping mattress will lie between the participant and the surface assessed to generate a pressure map.

Following completion of data collection, data will be analysed and any areas of potential pressure damage vulnerability will be identified.

ELIGIBILITY:
Inclusion criteria:

• Subjects will be individuals aged 18 and over, with good command of spoken and written English, full mobility, and the capacity to give informed, written consent. Provided there is no impairment to mobility, there is no upper age limit to participation.

Exclusion criteria:

* Inability to provide informed written consent
* Having a BMI that falls outside of the stated ranges for the study (<19)
* Any significant impairment to mobility, for whatever reason, that prevents the patient from getting in and out of bed unaided, walking 100 metres unaided, or climbing a flight of stairs unaided.
* Patients who lack sufficient command of written and spoken English to allow them to give written informed consent take part.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in the study will be adults with full mobility, with the capacity to give informed written consent. We will recruit a group of volunteers in order represent a variety of BMIs, in an attempt to gain a sample of the BMIs found in the population.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
PRESSURE AREA DISTRIBUTION ON A VARIETY OF CLINICAL SURFACES IN A GROUP OF 51 VOLUNTEERS | 125 minutes
  Establish the pressure distributions of current patient surfaces in use, for a variety of different sized patients, to identify any points in the patient's journey when they are at risk of developing pressure damage.

SECONDARY OUTCOMES:
PRESSURE AREA DISTRIBUTION ON A VARIETY OF CLINICAL SURFACES IN A GROUP OF 51 VOLUNTEERS | 125 minutes
  Gain information to allow calculation of a sample size for a definitive study.

CONTACTS AND LOCATIONS:
Locations (1):
- Brighton and Sussex University Hospitals NHS Trust, Brighton, East Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The authors plan to disseminate the findings of this study by publishing in the academic literature.

REFERENCES:
- [Background] Bennett G, Dealey C, Posnett J. The cost of pressure ulcers in the UK. Age Ageing. 2004 May;33(3):230-5. doi: 10.1093/ageing/afh086. PMID 15082426
- [Background] Chen HL, Chen XY, Wu J. The incidence of pressure ulcers in surgical patients of the last 5 years: a systematic review. Wounds. 2012 Sep;24(9):234-41. PMID 25874704
- [Background] Dealey C, Posnett J, Walker A. The cost of pressure ulcers in the United Kingdom. J Wound Care. 2012 Jun;21(6):261-2, 264, 266. doi: 10.12968/jowc.2012.21.6.261. PMID 22886290
- [Background] DOWNIE F, GUY H, GILROY P, ROYALL D, DAVIES S. Are 95% of hospital-acquired pressure ulcers avoidable?. Wounds UK. 2013 Sep 1;9(3).
- [Background] Hibbs P. The economic benefits of a prevention plan for pressure sores. In4th National Pressure Sore Symposium, Bath 1988 Apr (Vol. 20).
- [Background] McInnes E, Jammali-Blasi A, Bell-Syer S, Dumville J, Cullum N. Preventing pressure ulcers--Are pressure-redistributing support surfaces effective? A Cochrane systematic review and meta-analysis. Int J Nurs Stud. 2012 Mar;49(3):345-59. doi: 10.1016/j.ijnurstu.2011.10.014. Epub 2011 Nov 20. PMID 22104042
- [Background] National Pressure Ulcer Advisory Panel, European Pressure Ulcer Advisory Panel and Pan Pacific Pressure Injury Alliance. Prevention and Treatment of Pressure Ulcers: Quick Reference Guide. Emily Haesler (Ed.). Cambridge Media: Perth, Australia; 2014.